CLINICAL TRIAL: NCT01497639
Title: Comparison of the Efficacy of Double Monopolar Versus Interleaving Stimulation Modes for the Deep Brain Stimulation Treatment of Primary Generalized or Segmental Dystonia
Brief Title: Comparison of the Efficacy of Double Monopolar Versus Interleaving Stimulation Modes for Pallidal Deep Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Dr. Norbert Kovacs, Associate professor, specialist in neurology and movement disorders, Department of Neurology, University of Pecs
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 760906
Record Dates: First submitted 2011-12-14; First posted 2011-12-22 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Primary Dystonia
Keywords: dystonia; pallidal stimulation; deep brain stimulation; deep brain stimulation of GPi; GPi; interleaving stimulation
MeSH Terms: conditions — Dystonic Disorders; Dystonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Process 1 (Active Comparator): * Visit 1: Baseline evaluation (maximum 1 week before operation)
  * Visit 2: Testing of electrodes and subsequent initiation of interleaving stimulation mode (4th postoperative week).
  * Visit 3 Evaluation and cross-over to double-monopolar stimulation mode (16th postoperative week).
  * Visit 4 Final evaluation. (28th postoperative week).
  Interventions: Device: Interleaving stimulation mode (Medtronic); Device: Double monopolar stimulation mode (Medtronic)
- Process 2 (Active Comparator): * Visit 1: Baseline evaluation (maximum 1 week before operation)
  * Visit 2: Testing of electrodes and subsequent initiation of double-monopolar stimulation mode (4th postoperative week).
  * Visit 3 Evaluation and cross-over to interleaving stimulation mode (16th postoperative week).
  * Visit 4 Final evaluation. (28th postoperative week).
  Interventions: Device: Interleaving stimulation mode (Medtronic); Device: Double monopolar stimulation mode (Medtronic)

INTERVENTIONS:
Device: Interleaving stimulation mode (Medtronic) — Interleaving stimulation mode with constant frequency (125 Hz) and pulse-width (120us)parameters 'Interleavingr stimulation mode (Medtronic)'
  Other Names: Medtronic Activa RC Interleaving Stimulation Mode
Device: Double monopolar stimulation mode (Medtronic) — Double monopolar stimulation mode with constant frequency (125 Hz) and pulse-width (120us)parameters 'Double monopolar stimulation mode (Medtronic)'
  Other Names: Medtronic Activa RC Double Monopolar Stimulation Mode

SUMMARY:
The aim of the study is to compare the efficacy and the safety profile of the newly introduced interleaving stimulation mode to those of the standard double monopolar stimulation mode during pallidal deep brain stimulation of primary generalized or segmental dystonia.

DETAILED DESCRIPTION:
Background:

For the treatment of drug-refractory dystonia, bilateral pallidal deep brain stimulation (GPi-DBS) is proven to be an efficient option. On average, 40-55% improvement on dystonia rating scales (DRS) could be achieved according to the results of multicenter trials lasting for years. However, a considerable portion (10-25%) of the patients experience minimal alleviation despite of good electrode placement. These patients can be regarded as non-responders to GPi-DBS defined as having either limited improvement (< 25% on DRS) or worsening. Besides adjusting the amplitude, frequency or pulse-width of stimulation, one can change the electrode configuration from the commonly applied single monopolar stimulation mode (one contact on the electrode is negative) to either double monopolar stimulation (two -usually adjacent- negative contacts on the electrode are stimulated with same amplitude and pulse-width values) or bipolar stimulation mode (one contact on the electrode is positive) in case of unsatisfactory outcomes. Although these techniques had been utilized in multicenter trials, non-responsiveness to GPi-DBS did occur. Recently the investigators have reported in the Movement Disorders that the newly introduced interleaving stimulation mode was superior to single or double monopolar stimulation in four patients who had initially (6-12 months after implantation) limited response to GPi DBS.

Aims of the study:

To systematically compare the efficacy and the side-effect profile of double monopolar stimulation mode to those of interleaving stimulation mode in a prospective, randomized, double-blind, and cross-over study.

Methods:

The investigators would enroll 20-25 patients with drug refractory segmental or generalized primary dystonia undergoing bilateral GPi-DBS implantation within a 2-3 year time frame. The inclusion and exclusion criteria would follow those of the study of Kupsch et al.

ELIGIBILITY:
Inclusion Criteria:

* ages of 7 and 75 years
* marked disability owing to primary generalized or segmental dystonia, despite optimal pharmacologic treatment
* disease duration of at least 5 years.

Exclusion Criteria:

* previous brain surgery;
* cognitive impairment (< 120 points on the Mattis Dementia Rating Scale)
* moderate-to-severe depression (> 25 points on the Beck Depression Inventory)
* marked brain atrophy as detected by magnetic resonance imaging
* other medical or psychiatric coexisting disorders that could increase the surgical risk or interfere with completion of the trial

Ages: 7 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
Differences in severity of dystonia | 7 months
  Differences in severity of dystonia measured by Burke-Fahn-Marsden Dystonia Rating Scale

SECONDARY OUTCOMES:
Number of treatment responders after three months deep brain stimulation | 7 months
  Differences in number of treatment responders (at least 25% improvement on Burke-Fahn-Marsden Dystonia Rating Scale compared to baseline)
Health-related quality of life after three months deep brain stimulation | 7 months
  Differences in health-related quality of life measured by EQ-5D and SF-36 scales
Side-effect profile after three months deep brain stimulation | 7 months
  Differences in side-effect profile measured by stuctured deep brain stimulation-related side-effect questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Kovacs, MD, PhD, Principal Investigator — Associate professor, Department of Neurology, University of Pecs
Locations (1):
- Department of Neurology, University of Pécs, Pécs, Baranya, Hungary

REFERENCES:
- [Background] Kupsch A, Benecke R, Muller J, Trottenberg T, Schneider GH, Poewe W, Eisner W, Wolters A, Muller JU, Deuschl G, Pinsker MO, Skogseid IM, Roeste GK, Vollmer-Haase J, Brentrup A, Krause M, Tronnier V, Schnitzler A, Voges J, Nikkhah G, Vesper J, Naumann M, Volkmann J; Deep-Brain Stimulation for Dystonia Study Group. Pallidal deep-brain stimulation in primary generalized or segmental dystonia. N Engl J Med. 2006 Nov 9;355(19):1978-90. doi: 10.1056/NEJMoa063618. PMID 17093249
- [Background] Vidailhet M, Vercueil L, Houeto JL, Krystkowiak P, Benabid AL, Cornu P, Lagrange C, Tezenas du Montcel S, Dormont D, Grand S, Blond S, Detante O, Pillon B, Ardouin C, Agid Y, Destee A, Pollak P; French Stimulation du Pallidum Interne dans la Dystonie (SPIDY) Study Group. Bilateral deep-brain stimulation of the globus pallidus in primary generalized dystonia. N Engl J Med. 2005 Feb 3;352(5):459-67. doi: 10.1056/NEJMoa042187. PMID 15689584
- [Background] Valldeoriola F, Regidor I, Minguez-Castellanos A, Lezcano E, Garcia-Ruiz P, Rojo A, Salvador A, Castro A, Grandas F, Kulisevsky J, Marti MJ, Martinez-Martin P, Relova L, Rumia J, Camara A, Burguera JA, Linazasoro G, de Val JL, Obeso J, Rodriguez-Oroz MC, Tolosa E; Grupo ESpanol para el EStudio de la EStimulacion PALidal en la DIStonia. Efficacy and safety of pallidal stimulation in primary dystonia: results of the Spanish multicentric study. J Neurol Neurosurg Psychiatry. 2010 Jan;81(1):65-9. doi: 10.1136/jnnp.2009.174342. Epub 2009 Sep 10. PMID 19744963
- [Background] Vidailhet M, Vercueil L, Houeto JL, Krystkowiak P, Lagrange C, Yelnik J, Bardinet E, Benabid AL, Navarro S, Dormont D, Grand S, Blond S, Ardouin C, Pillon B, Dujardin K, Hahn-Barma V, Agid Y, Destee A, Pollak P; French SPIDY Study Group. Bilateral, pallidal, deep-brain stimulation in primary generalised dystonia: a prospective 3 year follow-up study. Lancet Neurol. 2007 Mar;6(3):223-9. doi: 10.1016/S1474-4422(07)70035-2. PMID 17303528
- [Background] Kupsch A, Tagliati M, Vidailhet M, Aziz T, Krack P, Moro E, Krauss JK. Early postoperative management of DBS in dystonia: programming, response to stimulation, adverse events, medication changes, evaluations, and troubleshooting. Mov Disord. 2011 Jun;26 Suppl 1:S37-53. doi: 10.1002/mds.23624. PMID 21692111
- [Background] Kovacs N, Janszky J, Nagy F, Balas I. Changing to interleaving stimulation might improve dystonia in cases not responding to pallidal stimulation. Mov Disord. 2012 Jan;27(1):163-5. doi: 10.1002/mds.23962. Epub 2011 Sep 28. No abstract available. PMID 21956680
- [Background] Tagliati M, Krack P, Volkmann J, Aziz T, Krauss JK, Kupsch A, Vidailhet AM. Long-Term management of DBS in dystonia: response to stimulation, adverse events, battery changes, and special considerations. Mov Disord. 2011 Jun;26 Suppl 1:S54-62. doi: 10.1002/mds.23535. PMID 21692113